CLINICAL TRIAL: NCT01876355
Title: The Effect of Clonidine-enhanced Sedation on Delirium in Ventilated Critically Ill Patients CATAPRES (Confusion and Alpha-Two Agonist Prescription Randomised Efficacy Study)
Brief Title: The Effect of Clonidine-enhanced Sedation on Delirium in Ventilated Critically Ill Patients
Acronym: CATAPRES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Deventer Ziekenhuis (Other)
Responsible Party: Principal Investigator, Marieke Zeeman, Principal Investigator, Deventer Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cat1.1
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Delirium
Keywords: Delirium, clonidine, ICU, sedation
MeSH Terms: conditions — Delirium | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clonidine (Experimental)
  Interventions: Drug: Clonidine
- Sodium chloride (Placebo Comparator)
  Interventions: Drug: SodiumChloride

INTERVENTIONS:
Drug: Clonidine — o The concentration of clonidine in the solution is 12.5 µg/ml. Continuous iv infusion of 0.02 ml/kg/h results in a dosage of 0.25 µg/kg/h. The maximum dosage achieved is 25 µg/h. The total amount of clonidine given to a person with a body weight 100 kg or more will be 600 µg a day. Since the doses chosen are in the low range, there will be no dosage adjustment for renal- or liver failure.
  Other Names: Catapressan
  Arms: Clonidine
Drug: SodiumChloride — Placebo. Pharmaceutical form: Injection. Route of administration: Intravenous use.
  Other Names: Placebo
  Arms: Sodium chloride

SUMMARY:
Rationale: Delirium is highly prevalent in the ICU. GABA-ergic anaesthetics may provoke delirium. Alpha-2-adrenergic agonists may lead to a reduction of the total amount of GABA-ergic anaesthetics and reduction of delirium. There are no large studies proving that this therapy is effective and safe.

Objective: The objective of this study is to compare the effect of clonidine with placebo on the occurrence and duration of delirium in mechanically ventilated ICU patients.

Study design: Prospective randomised double-blind placebo controlled intervention study in 115 patients.

Study population: All patients >18 years old, intubated mechanically ventilated and sedated at inclusion.

Intervention: Clonidine infusion of 0,25 mcg/kg/h added to the standard sedation regimen. Comparison: NaCl 0,9 % infusion as placebo.

Main study parameters/endpoints: The main study parameter is the total number of awake and delirium-free observation periods the first 7 days after randomisation. An observation period is a nursing shift of 8 hours.

DETAILED DESCRIPTION:
Rationale: Delirium is highly prevalent in the ICU. It may cause significant morbidity and mortality. One of the factors that may provoke a delirium is the use of GABA-ergic anaesthetics. Recent studies have shown that sedation with alpha-2-adrenergic agonists may lead to a reduction of the total amount of GABA-ergic anaesthetics and reduction of delirium. In clinical practice the alpha-2-adrenergic agent clonidine is used as an add-on sedative in mechanically ventilated patients who suffer from delirium, but there are no large studies proving that this therapy is effective and safe.

Objective: The objective of this study is to compare the effect of clonidine with placebo on the occurrence and duration of delirium in mechanically ventilated ICU patients.

Study design: Prospective randomised double-blind placebo controlled intervention study in 115 patients.

Study population: All patients >18 years old, intubated mechanically ventilated and sedated at inclusion.

Intervention: Clonidine infusion of 0,25 mcg/kg/h added to the standard sedation regimen. Comparison: NaCl 0,9 % infusion as placebo.

Main study parameters/endpoints: The main study parameter is the total number of awake and delirium-free observation periods the first 7 days after randomisation. An observation period is a nursing shift of 8 hours.. A delirium-free period is a shift in which the CAM-ICU score is negative.

Secondary endpoints: RASS sedation score, total number of delirium positive observation periods, total amount of sedatives, analgesics and antipsychotics used, organ failure score, ventilation and sedation free days at day 30, mortality.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden associated with participation is minimal. All blood samples, CAM-ICU scores and physical examinations required for the study are routine daily practice on the ICU. Adding clonidine for sedation of critically ill patients is common practice in many ICU's in the Netherlands.. Its use is also suggested in the NVIC guideline delirium on the ICU. It is however an off-label treatment. The major side effects of the study medication clonidine are hypertension, hypotension and bradycardia. Smaller studies have shown that these side effects are comparable to midazolam. Hypotension is a phenomenon that occurs very often in ICU patients, and is caused by different conditions, not only by the use of sedative medication. The benefit of participation is the possibility to reduce the period of delirium during ICU stay. Because of the widely off label use of clonidine in sedated and ventilated critically ill ICU patients this study is relevant to test the hypothesis that sedation with clonidine leads to a lower incidence and shorter duration of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated, at the start of the study medication.
* Age > 18 years

Exclusion Criteria:

* Severe neurotrauma/CVA
* Severe dementia
* Inability to speak Dutch or English
* The use of clonidine during the 96 hours before the start of the study.
* Bradycardia (<50/min)
* Severe hypotension (MAP < 65 after volume resuscitation and two vasopressors)
* Pregnancy
* Epilepsy
* Known clonidine intolerance
* Liver cirrhosis (Child-Pugh Class C)
* Recent and acute myocardial infarction
* Severe heart failure (LVEF<30%)
* Second or third degree AV block
* Renal insufficiency requiring intermittent haemodialysis (CVVH is permitted)
* Expected transfer to another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
CAM-ICU (Confusion Assessment Method for the Intesive Care Unit) | 7 days
  The total amount of delirium-free periods during 7 days after randomisation and start of the study medication. An observation period is a period of 8 hours, coinciding with one nursing shift. A delirium-free period is a shift in which the delirium score is negative.

SECONDARY OUTCOMES:
Signs of agitation | 7 days
  Signs of agitation (for example self removed catheter).
Opiate use | 7 days
Sedative use | 7 days
Anti-psychotic use | 7 days
Ventilation free days | 7 days
Sedation free days | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: H.L.A. van den Oever, Principal Investigator — Deventer Ziekenhuis
Locations (1):
- Deventer Hospital, Deventer, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No